CLINICAL TRIAL: NCT04454008
Title: Executive Functioning Family Training for Preschool Children With Attention Deficit Hyperactivity Disorder - a Randomized Controlled Study
Brief Title: RCT of EF Family Training for P ADHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-20-012
Record Dates: First submitted 2020-06-27; First posted 2020-07-01 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2020-05

CONDITIONS: ADHD
Keywords: ADHD; executive function; preschool; intervention; RCT
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Coal Tar

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The evaluator was unaware of the subjects' treatment status
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive 12 sessions of executive function family training, including executive function training for children and parenting guidance for parents.
  Interventions: Behavioral: executive function family training
- waiting (Active Comparator): The waiting group will receive routine clinical intervention, including health education, family support and guidance from outpatient clinic.
  Interventions: Behavioral: treat as usual

INTERVENTIONS:
Behavioral: executive function family training — Intervention programs include executive function training for children with ADHD and parenting guidance for parents
  Arms: Intervention
Behavioral: treat as usual — Outpatient routine health education, behavioral guidance and family support
  Arms: waiting

SUMMARY:
To explore the effect of executive function family training for preschool children with ADHD, providing early social psychological intervention for aiming the core impairments of ADHD.

DETAILED DESCRIPTION:
100 preschool children with ADHD will be randomly divided into the intervention group and the waiting group. The waiting group received regular clinical intervention, while the intervention group received 12-week training. The intervention program includes executive function training for ADHD children and parenting guidance for parents by two therapists respectively, which were carried out in two meeting rooms in Xinhua Hospital. Therapists are psychiatrists with a background in child psychiatry and psychotherapists with training in ADHD area. After 12 weeks, the improvement of ADHD core symptoms and executive function was compared.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria for preschool ADHD, based on the the DSM-5 criteria by the attending physician or above;
* Age 4 months 0 to 5 years 11 months;
* Total IQ is above 80 assessed by WPPSI.

Exclusion Criteria:

* Attention deficit disorders resulting from organic neurological diseases, extensive developmental disorders, mental retardation, childhood schizophrenia, mood disorders, epilepsy, and other organic diseases or other primary mental disorders;
* parent or guardian with a serious mental illness, such as schizophrenia, mood disorder (onset), etc., and Educational level is lower than junior middle school;
* Participants who failed to attend more than 80% of the intervention sessions (at least 9 sessions).

Ages: 48 Months to 71 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2020-12-06 (Actual); Primary Completion 2023-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
ADHD core symptoms | 12 weeks after baseline
  ADHD core symptoms are assessed by Swanson, Nolan, and Pelham Rating Scale (SNAP), with the score ranged from 0-54 (the higher the socre, the worse the symptoms)

SECONDARY OUTCOMES:
Executive function-Inhibition | 12 weeks after baseline
  The executive function inhibition is assessed by NEPSY-II task Status (ST) with the higher the score is, the better the function.
Executive function-working memory | 12 weeks after baseline
  The executive function working memory is assessed by NEPSY-II task memory design (MD) with the higher the score is, the better the function.

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Zhang, Doctor, Study Director — Director of department of psychology, xinhua hospital
Locations (1):
- Xinhua Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No